CLINICAL TRIAL: NCT06759701
Title: Pre-Surgical Tirzepatide-Assisted Weight Loss in Overweight and Obese Men With Intermediate Risk Prostate Cancer: A Pilot Feasibility Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-1496; NCI-2024-10696 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-12-29; First posted 2025-01-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Diabetes; Prostate Cancer
MeSH Terms: conditions — Diabetes Mellitus; Prostatic Neoplasms | interventions — Tirzepatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tirzepatide (Experimental)
  Interventions: Drug: Tirzepatide

INTERVENTIONS:
Drug: Tirzepatide — Participants will perform weekly self-injection of tirzepatide as standard of care, following manufacturer instructions

SUMMARY:
The goal of this clinical research study is to determine how well a tirzepatide-assisted weight loss program works before a prostatectomy in patients with intermediate risk prostate cancer

DETAILED DESCRIPTION:
Primary Objectives:

To determine the feasibility of a tirzepatide-assisted weight loss program prior to radical prostatectomy in a group of men diagnosed with intermediate risk prostate cancer, defined based on the following process measures:

Enrollment (completion of 30 patient accrual within 2 years) Retention (completion of the study through the day of surgery, with ≥90% defined as successful) Adherence (the percentage of completed study sessions and clinic visits, with ≥70% considered successful).

Secondary Objectives:

1. Determine differences in plasma and tumor sphingolipids following tirzepatide-based intervention
2. Determine differences in markers of insulin and insulin signaling following tirzepatide-based intervention
3. Determine differences in prostate, plasma and periprostatic fat inflammatory signaling following tirzepatide-based intervention
4. Determine differences in tumor proliferation following tirzepatide-based intervention, including when stratified by obesity- and prostate cancer-associated SNPs and GLP-1 expression.
5. Determine differences in ASCVD risk factors following tirzepatide-based intervention.
6. Determine differences in other markers of cardiovascular risk.
7. Determine changes in body scan as measured by DEXA scan after tirzepatide-based intervention
8. Determine change in body weight following tirzepatide-based intervention.
9. Determine changes in gut microbiome alpha and beta diversity following tirzepatide-based intervention.
10. Determine rates of biochemical recurrence, receipt of salvage radiation therapy, and receipt of androgen deprivation therapy, stratified by prostatectomy pathology, after tirzepatidebased intervention

Correlative Outcomes Cardiovascular, Surgical, and Patient-Related Outcomes Outcome Measure Outcome Measure Difference in plasma sphingolipids Change in plasma sphingolipid signature from baseline to pre-surgery within patients Difference in ASCVD risk factor score Change in the Metabolic Syndrome Severity Score (MetSSS)32

Difference in insulin signaling Compare change in fasting insulin, IGFBP-3, IGF-1 and C-peptide within patients Difference other markers of cardiovascular disease risk Between-group difference hsCRP, YKL-40, ICAM-1, E-selectin, leptin, and lipoproteins (e.g. LDL, LP(a)) Difference in tumor and periprostatic fat inflammatory markers Tumor and peri-prostatic fat inflammatory mRNA levels (CXCL12, CXCL1, CCR7 and IL-6, TNF-α) Change is DEXA-defined body composition measures Change in body fat percent, appendicular lean mass index, and other indices Compare tumor ki67 and other relevant proteins stratified by tumor GLP-1 receptor expression and Decipher score Spearman correlation of tumor ki67 change with GLP-1 receptor density (based on IHC). Analyses stratified by Decipher and other groups, as well. Change in body weight Change in the absolute body weight

Determine differences in tumor proliferation stratified by germline obesity- and prostate cancer-associated germline SNPs Stratified analysis of ki67 expression based on germline genotype at rs12529, rs6161, rs523349, and rs1047303.

Determine changes in the gut microbiome with use of GLP-1 assisted weigh loss Established measures of alpha and beta diversity of microbial species

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate that is localized (no metastatic lesions or concerning lymph nodes 1cm or greater) based on prostate MRI and meets NCCN intermediate risk criteria (as follows):

  * Clinical T2b-T2c or lower disease
  * Gleason Grade group 2 or 3 on biopsy
  * PSA ≤20 ng/mL
  * Desires radical prostatectomy (open or robotic) for prostate cancer management and is a surgical candidate as determined by the treating urologic oncologist
* Adult men >30 and < 75 years old
* Currently diagnosed with Diabetes Mellitus and meet one of the following criteria for overweight or obesity:

  * Body Mass Index (BMI) greater than or equal to 27 kg/m2
  * Waist circumference (> 40 inches) -or-
* Currently have a BMI greater or equal to 30 kg/m2 -or-
* Currently have a BMI greater or equal to 27 kg/m2 with at least one weight-related condition, defined as one or more of the following:

  * Hypertension: treated or with systolic blood pressure (SBP) ≥130 mmHg or diastolic blood pressure ≥80 mmHg
  * Dyslipidemia: treated or with low-density lipoprotein (LDL) ≥160 mg/dL (4.1 mmol/L) or triglycerides ≥150 mg/dL (1.7 mmol/L), or high-density lipoprotein (HDL) <40mg/dL (1.0 mmol/L)
  * Obstructive sleep apnea
  * Cardiovascular disease (for example, ischemic cardiovascular disease, New York Heart Association (NYHA) Functional Class I-III heart failure)

Exclusion Criteria:

* Prostate cancer that meets factors as part of NCCN high and very high-risk criteria (as follows):

  * pT3a or higher disease
  * Grade group 4 or 5 adenocarcinoma of prostate
* Presence of metastatic disease on imaging
* A history of intentional or unintentional weight loss of more than 5kg within 90 days of screening
* Any prior androgen deprivation, chemotherapy, surgery, or radiation for PCa
* Previous or planned surgical treatment for obesity or use of a medication that promotes weight loss within 90 days before screening
* Have renal impairment measured as estimated glomerular filtration rate (eGFR) <30 as determine using standard MD Anderson laboratory measures
* Have a known clinically significant gastric emptying abnormality (for example, severe diabetic gastroparesis or gastric outlet obstruction) or chronically take drugs that directly affect GI motility
* Have had a history of chronic or acute pancreatitis
* Have a history of significant active or unstable Major Depressive Disorder (MDD) or other severe psychiatric disorder (for example, schizophrenia, bipolar disorder, or other serious mood or anxiety disorder) within the last 2 years

  * Note: Patients with MDD or generalized anxiety disorder whose disease state is considered stable and expected to remain stable throughout the course of the study, in the opinion of the investigator, may be considered for inclusion if they are not on excluded medications
* Have any of the following cardiovascular conditions within 3 months prior to study enrollment: acute myocardial infarction (MI), cerebrovascular accident (stroke), unstable angina, or hospitalization due to congestive heart failure (CHF)
* Have NYHA Functional Classification IV CHF
* Have acute or chronic hepatitis, signs, and symptoms of any other liver disease other than nonalcoholic fatty liver disease, or any of the following, as determined by the central laboratory during screening: - alanine aminotransferase (ALT) level >3.0X the upper limit of normal (ULN) for the reference range or - alkaline phosphatase (ALP) level >1.5X the ULN for the reference range or - total bilirubin level >1.2X the ULN for the reference range (except for cases of known Gilbert's Syndrome) Note: Participants with nonalcoholic fatty liver disease are eligible to participate in this trial if their ALT level is ≤3.0X the ULN for the reference range
* Have a family or personal history of medullary thyroid carcinoma (MTC) or Multiple Endocrine Neoplasia (MEN) Syndrome type 2
* Have a history of an active or untreated malignancy or are in remission from a clinically significant malignancy (other than basal- or squamous-cell skin cancer, in situ carcinomas of the cervix), other than prostate cancer, for less than 5 years
* Have any other condition not listed in this section (for example, hypersensitivity or intolerance) that is a contraindication to GLP-1R agonists
* Have a history of any other condition (such as known drug or alcohol abuse, diagnosed eating disorder, or other psychiatric disorder) that, in the opinion of the investigator, may preclude the participant from following and completing the protocol
* Have history of use of marijuana within 3 months of enrollment and unwillingness to abstain from marijuana use during the trial. Participants should also refrain from use of cannabidiol oil for the duration of the study
* Have had a transplanted organ (corneal transplants [keratoplasty] allowed) or awaiting an organ transplant.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Justin Gregg, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M. D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org